CLINICAL TRIAL: NCT03952754
Title: Effect of an Integrated Nutrition-math Curriculum to Improve Food-purchasing Behavior of Children
Brief Title: Effect of Hip Hop Nutrition-Math Curriculum
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative changes
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Olajide Williams, Associate Professor of Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAR5173; 5R01NR017571 (NIH)
Record Dates: First submitted 2019-05-11; First posted 2019-05-16 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Health Behavior
Keywords: Nutrition; Health; School Children
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 2: Hip Hop Nutrition-Math Curriculum (Experimental): The intervention group will receive an tailored program for ten weeks, meeting twice a week.
  Interventions: Behavioral: Hip Hop Nutrition-Math Curriculum
- Group 1: Food Explorers Program (Active Comparator): The control group will receive the usual care for nutrition program provided by the schools, called Food Explorers. The group will also be conducted ten weeks, meeting twice a week.
  Interventions: Behavioral: Food Explorers Program

INTERVENTIONS:
Behavioral: Hip Hop Nutrition-Math Curriculum — This program teaches children skills needed to understand restaurant-menu boards, how to make healthy food choices, while reinforcing the common core math concepts they are learning in school. The program consists of: 2 lessons a week, of about 1 hour each lesson, for a total of 20 lessons.
  Other Names: Hip Hop Nutrition math-based education program
  Arms: Group 2: Hip Hop Nutrition-Math Curriculum
Behavioral: Food Explorers Program — After-school program Food Explorers will represent "Usual Care". This program comprises food and exploration activities, familiarizing children with diverse foods, nutrition concepts, tasty recipes and physical activity.
  Other Names: Food Explorers Curriculum
  Arms: Group 1: Food Explorers Program

SUMMARY:
This study is testing the efficacy of the integrative approach to:

1. teach 5th grade children menu board calorie literacy as measured by our novel recently validated menu board calorie literacy (MBCL) instrument;
2. provide strategies designed to improve food purchasing behaviors; and
3. facilitate the transmission of core lesson messages from children to parents via a procedure that we have termed "Child Mediated Health Communication (CMHC)".

DETAILED DESCRIPTION:
Data show that nearly 25% of children aged four to eight years consumed fast food on a typical day. These trends in fast food consumption are more acute among low-income urban dwellers where higher rates of overweight and childhood obesity are seen. This has led to a focus on providing fast food consumers with point-of-purchase nutrition information, such as the calorie posting mandates, in the hopes that these decision cues will help consumers make better informed dietary decisions. Most children chose their own meals at the point-of-purchase. It is clear that additional strategies are needed to encourage the point-of-purchase use of calorie postings, however available studies provide little insight into best practices or the types of approaches needed.

It is with this in mind that the investigator developed a school-based approach to improve point-of purchase use of calorie postings, by creating a novel intervention that targets menu board calorie literacy as a means of improving food-purchasing behaviors.

Hip Hop Nutrition-Math Curriculum is a novel behaviorally focused multimedia, musical school health rap toolkit that targets what we refer to as menu board calorie literacy. 4th grade common core math standards are integrated into the program in a manner that incorporates evidence-based nutrition education recommendations by the Institute of Medicine and the Centers for Disease Control and Prevention (CDC).

The investigator proposes to test the efficacy of the integrative approach on food purchasing behaviors of children in an adequately powered, controlled trial. The investigator will test the intervention in the after-school setting among economically disadvantaged children and incorporate parental engagement in our outcome evaluations. There is a partnership with New York City's largest after-school program vendor, New York Edge (formerly called Sports and Arts in Schools foundation/SASF), for the implementation of this study.

The goal of a health literacy intervention is to improve health decision-making and/or behavior. For this reason, the investigator will measure both menu board calorie literacy and food choice behavior at a point-of-purchase.

ELIGIBILITY:
Inclusion Criteria:

* 5th grade student participating in the New York Edge after school program

Exclusion Criteria:

* Absence of Internet access at home
* No working phone line
* Major psychiatric disability or medical condition that may affect participation (e.g., psychotic illness, terminal illness)
* Non-English speaking students

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 560 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of students with positive behavior change at Food Sales | Within Year5 of the study
  Students will be tracked on the food purchases they make at "Food Sales" conducted through study.
  Each child will be given an identifiable food voucher for use at the Food Sale. However, point-of-purchase behaviors will be assessed with the children unaware that their food choices being tracked. The food categories range from low calorie/nutrient to high.
  A change from a purchase of a high-calorie/nutrient item to a low-calorie/nutrient item will indicate a positive behavior change.

SECONDARY OUTCOMES:
Menu Board Calorie Literacy Score | Baseline, Post-Intervention (approximately 10 Weeks), 3-Month Follow Up
  Content knowledge of students will be assessed by the total number of correct responses on the survey measures.
Parental Nutritional Knowledge Score | Baseline, Post-Intervention (approximately 10 Weeks), 3-Month Follow Up
  Nutrition knowledge score will be assessed using a 7-item questionnaire at Baseline, Immediately post intervention, and at 3-months post intervention. Changes in the composite score will be analyzed across each of the test sequences range of 0 - 7, with higher scores representing greater nutrition knowledge.

OTHER OUTCOMES:
Exploratory Outcome Measures: BMI Percentiles | Baseline, Post-Intervention (approximately 10 Weeks), 3-Month Follow Up
  The change in BMI percentiles from a high-index to low-index will indicate a change in BMI and program impact.

CONTACTS AND LOCATIONS:
Overall Officials: Olajide A. Williams, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No